CLINICAL TRIAL: NCT06973330
Title: Sintilimab Plus Apatinib and SOX as First-line Treatment in Patients With AFP Gastric or Gastroesophageal Junction Adenocarcinoma: a Single-arm, Multi-center, Phase II Trial
Brief Title: Sintilimab Plus Apatinib and SOX as First-line Treatment in Patients With AFP Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Provincial Cancer Hospital (Other)
Responsible Party: Principal Investigator, Juan Cai, chief physician, Anhui Provincial Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-Ethic-156
Record Dates: First submitted 2025-04-18; First posted 2025-05-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-01

CONDITIONS: AFP Gastric or Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — sintilimab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Drug: Apatinib and Sintilimab SOX regimen combined with Sintilimab and Apatinib
  Interventions: Drug: SOX regimen combined with Sintilimab and Apatinib

INTERVENTIONS:
Drug: SOX regimen combined with Sintilimab and Apatinib — Patients who met the inclusion criteria were treated with SOX regimen combined with Sintilimab plus Apatinib every 3 weeks(4 cycles) followed by sintilimab+apatinib until disease progression or intolerable adverse reactions or death(up to 24 months).

SUMMARY:
This is a multi-center, prospective, open label phase II study evaluating the safety and efficacy of standard first-line chemotherapy SOX regimen combined with Sintilimab (anti-PD-1 antibody) and Apatinib in the treatment of advanced AFP-positive gastric cancer. This study was conducted in the Department of Anhui Provincial Cancer Hospital. In this study, patients with AFP-positive and HER-2-negative advanced gastric cancer who had not received palliative systematic treatment in the past will be enrolled. Patients who met the inclusion criteria were treated with SOX regimen combined with Sintilimab plus Apatinib every 3 weeks(4 cycles) followed by sintilimab+apatinib until disease progression or intolerable adverse reactions or death(up to 24 months).Patients received regular and periodic reviews, with imaging evaluations every 6 weeks. Safety will be evaluated by AE and laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years old;
2. Patients with advanced / metastatic gastric cancer diagnosed by histopathology, without liver like differentiation, HER-2 negative, serum AFP ≥ 2xULN or AFP positive by the IHC staining;
3. No previous palliative systemic treatment;
4. There are measurable metastatic lesions according to RECIST version 1.1;
5. ECOG physical status score is 0 or 1；
6. Normal organ function: Neutrophil count ≥ 1.2 × 109/L, Platelet count ≥ 100 × 109/L, Hemoglobin (HB) ≥ 80g/L, Total bilirubin ≤ 1.5mg/dl, AST and ALT ≤ 100 IU/L. If the abnormal liver function is due to liver metastasis, AST and ALT should be ≤ 200 IU/L, Creatinine ≤ 1.5 times* upper limit of normal, International standardization ratio (INR) ≤ 1.5;
7. Urinary protein: meet one of the following conditions Urinary protein (test paper method) is 2 + or less, Urinary protein/creatinine (UPC) ratio < 3.5, Determination of 24-hour urinary protein, urinary protein ≤ 3500mg;
8. Before receiving treatment, the patient has recovered the adverse events related to chemotherapy, radiotherapy and surgery to grade 1 or below (CTCAE 5.0);
9. For women with fertility potential with negative pregnancy test within 14 days before enrollment, male and female patients should agree to use appropriate contraceptive methods from the beginning of the first treatment to 120 days after the last treatment;
10. Patients who can take oral drugs;
11. Signed the informed consent.

Exclusion Criteria:

1. Patients who received surgery and radiotherapy within 2 weeks before enrollment;
2. Patients who have previously been treated with Apatinib or any anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs;
3. Patients with uncontrollable hypertension (systolic blood pressure ≥ 160mmHg and diastolic blood pressure ≥ 90mmHg);
4. Patients with acute coronary syndrome (including myocardial infarction and unstable angina) who had undergone coronary angioplasty within 6 months before enrollment;
5. Patients with symptomatic brain metastases;
6. Patients with New York Heart Association (NYHA) grade II or above congestive heart failure or severe arrhythmia with severe cardiovascular damage in the past 6 months;
7. The patients had active malignancies in the past 24 months (except for melanoma in situ, basal cell carcinoma of the skin or squamous cell carcinoma or carcinoma in situ of the cervix) ;
8. The patients have severe (hospitalized) complications;
9. Patients with a history of gastrointestinal perforation and/or gastrointestinal fistula within 6 months before enrollment;
10. Patients with active hepatitis;
11. Patients with a history of human immunodeficiency virus (HIV) infection; 12. Patients with symptoms or signs of active interstitial pulmonary disease; 13. Patients with autoimmune diseases or a history of chronic or recurrent autoimmune diseases;

14. Patients who need systemic corticosteroids (excluding temporary use for testing, prophylactic administration of allergic reactions or reduction of swelling associated with radiotherapy) or immunosuppressants, or patients who receive such treatment within 14 days before enrollment; 15. The patient has a history of (non-infectious) pneumonia requiring steroids or has a current history of pneumonia; 16. Patients who received live vaccine < 30 days before starting trial drug treatment; The patient has serious non-healing wounds, ulcers or fractures; 17. Pregnant or lactating women; 18. The investigator determined that the patient is not suitable to be the subject of this trial; 19. Other circumstances that the investigator considers inappropriate to participate in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 24 months
  the rate of patients with PR and CR

SECONDARY OUTCOMES:
OS | 24 months
  The time from the beginning of treatment to the time when the patient dies from any cause
PFS | 24 months
  The time from the beginning of treatment to the time when the disease progresses or the patient dies from any cause

OTHER OUTCOMES:
AE | 24 months
  Safety will be evaluated by AE

IPD SHARING:
Plan to Share IPD: Undecided